CLINICAL TRIAL: NCT07077265
Title: Comparing Two Different Norepinephrine Infusion Rates for Prophylaxis Against Spinal-induced Hypotension in Elderly Patients Undergoing Hip Surgery: A Randomized Controlled Non-inferiority Trial
Brief Title: Comparing Two Different Norepinephrine Infusion Rates for Prophylaxis Against Spinal-induced Hypotension in Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-25-2024
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Spinal Aneshtesia; Hypotension After Spinal Anesthesia; Elderly (People Aged 65 or More)
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NE 0.1 mcg (Active Comparator): norepinephrine infusion rate of 0.1 mcg/kg/min
  Interventions: Drug: Norepinephrine (0.1 μg/kg/min)
- NE 0.07 mcg (Active Comparator): norepinephrine infusion rate of 0.07 mcg/kg/min
  Interventions: Drug: Norepinephrine (0.07 μg/kg/min)

INTERVENTIONS:
Drug: Norepinephrine (0.1 μg/kg/min) — The patients will receive norepinephrine infusion at a rate 1 mL/kg/hour of 6 mcg/mL solution.
  Arms: NE 0.1 mcg
Drug: Norepinephrine (0.07 μg/kg/min) — The patients will receive NE infusion at a rate 1 mL/kg/hour of 4.2 mcg/mL solution.
  Arms: NE 0.07 mcg

SUMMARY:
Hip surgery in the elderly is commonly performed under spinal anesthesia, which is associated with a lower risk of postoperative complications. However, this population is highly susceptible to postspinal hypotension-occurring in up to 69% of cases-which can compromise organ perfusion and increase the risk of organ failure and mortality. Vasodilation-induced hypotension is typically managed with vasopressors, and norepinephrine, with both α- and weak β-agonist activity, has recently been introduced as a prophylactic agent in this setting. Prior research demonstrated that a norepinephrine infusion at 0.1 mcg/kg/min effectively prevented hypotension in elderly patients undergoing hip arthroplasty, but only one dose was tested. Given findings from obstetric studies suggesting lower effective doses, the current study aims to determine whether a lower infusion rate (0.07 mcg/kg/min) is non-inferior to the higher dose in maintaining intraoperative blood pressure. Identifying the optimal dose is important for minimizing drug exposure while ensuring hemodynamic stability.

DETAILED DESCRIPTION:
Baseline preoperative blood pressure will be recorded in the supine position as average of 3 reading with difference less than 5 mmHg in the mean arterial pressure.

Inferior vena cava collapsibility will be used to assess the patient's intravascular volume status.

After induction of spinal anesthesia, patients will receive the vasopressor infusion according to the previous randomization All drug preparations will be done by a research assistant who will be responsible for opening the envelope and group assignment with no further involvement in the study.

Any episode of hypotension (defined as mean arterial pressure (MAP) < 70% of the baseline or MAP<65mmHg) will be managed by 5 mcg norepinephrine.

If bradycardia (defined as heart rate less than 50 bpm) with hypotension occurred, it will be manged with 9 mg ephedrine. If bradycardia occurred with hypertension (MAP increase 20% over the baseline) and persisted for more than one reading, the vasopressor infusion will be stopped.

If hypertension occurred (defined as increased mean arterial pressure by > 20% of the baseline reading), vasopressor infusion will be decreased by 50%. If hypertension persisted 2 minutes after reduction of the infusion, the vasopressor infusion will be stopped. The vasopressor will be returned to 50% of the starting dose if there was further decline in blood pressure.

The infusion will continue for 45 minutes after spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (>65)
* ASA I-II-III
* scheduled for hip surgery under spinal anesthesia

Exclusion Criteria:

* Contraindication of spinal anesthesia
* history of allergy to any of the study's drugs,
* Patients with cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias)
* patients with uncontrolled hypertension

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
mean arterial pressure | 0 min after spinal anesthesia till 46 min after spinal anesthesia
  average mean arterial pressure

SECONDARY OUTCOMES:
incidence of hypotension | 0 min after spinal anesthesia till 46 min after spinal anesthesia
  defined as mean MAP < 70% of the baseline or MAP<65mmHg
incidence of reactive hypertension | 0 min after spinal anesthesia till 46 min after spinal anesthesia
  defined as mean MAP > 120% of the baseline
incidence of bradycardia | 0 min after spinal anesthesia till 46 min after spinal anesthesia
  defined as heart rate <50 bpm

CONTACTS AND LOCATIONS:
Overall Officials: Maha Mostafa, MD, Principal Investigator — Cairo University Kasr Alainy Faculty of Medicine
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.